CLINICAL TRIAL: NCT06317727
Title: Pulsed Field Ablation of Colorectal Polyps
Acronym: PULSAR
Status: Not yet recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Mirai Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: IRAS 337105
Record Dates: First submitted 2024-02-22; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Colon Polyp
Keywords: Colorectal polyps; Irreversible electroporation; Endoscopic ablation
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsy specimen of the colorectal mucosa after the ablation therapy to determine residual or recurrent polyps
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulsed Field Ablation group: The EndoVE (Endoscopic vacuum electrode) is moved endoscopically into surface contact with the polyp. A vacuum is employed through the EndoVE as required to assist contact with the device. An electrical field depth of 8-10mm and surface area of 2cm3 is treated per pulse application. The electrical pulses are produced by an electroporation generator (ePORE device). Larger polyps will require multiple applications to ensure the full surface area has been treated. An overlap with previously pulsed areas is preferable to ensure all of the polyp tissue is ablated. The patient will then be transferred to the step-down ward to monitor for any adverse events before being discharged on the same day. The patient will be requested to attend the clinic for an endoscopy follow up at 4-6 weeks post EndoVE polyp treatment to investigate the response.
  Interventions: Device: Irreversible Electroporation using EndoVE(Endoscopic Vacuum Electrode) and electrical pulses generated using ePORE(electroporation device)

INTERVENTIONS:
Device: Irreversible Electroporation using EndoVE(Endoscopic Vacuum Electrode) and electrical pulses generated using ePORE(electroporation device) — The use of pulsed field ablation via irreversible electroporation delivered during flexible lower gastrointestinal endoscopy

SUMMARY:
The goal of this observational study is to learn about the role of electroporation (the use of small electric pulses applied to tissue) in the treatment (ablation) of colorectal polyps. The main questions to answer in this pilot phase of the study are:

1. The safety of pulsed field ablation (PFA) for the removal of colorectal polyps
2. The efficacy and feasibility of PFA in the treatment of colorectal polyps using metrics such as treatment coverage, treatment time, post treatment fibrosis, post treatment recurrence and patient satisfaction

DETAILED DESCRIPTION:
Colorectal cancer is the commonest cancer of the digestive tract, the second commonest cause of cancer deaths in the western hemisphere and the third commonest cancer in the United Kingdom. Most bowel cancers arise from precancerous growths called polyps. Prompt and effective treatment of these polyps can potentially prevent or cure bowel cancer at its earliest stages. King's College Hospital runs a special service dedicated to treating these lesions called the Special Polyps and Early Colorectal Cancer Service (SPECCS) using a variety of methods. These techniques usually involve removing the polyps through endoscopic resection. Other options include laparoscopic surgery, robotic surgery and rarely, open surgery. These modalities of treatments come with a number of risks, are highly invasive, require extensive skill and also have a long waiting list.

Endoscopic ablation with electroporation offers the potential of treating colorectal polyps in an easier, faster and less invasive manner. Electroporation uses small, high frequency, electric pulses, applied on the surface of tissues to temporarily open up pores in the outer wall of these cells. These pores, disrupts the structure of the abnormal cells and cause cell death via apoptosis. This approach has been used to treat frail patients with advanced colored cancer who cannot undergo more aggressive forms of treatment and it is postulated that this technology also has the ability to deal with colorectal polyps. This study is a pilot research involving a small number of patients with colorectal polyps who will be treated with electroporation given during colonoscopy.

Patients who participate in this study will be treated using endoscopic electroporation with the intent of ablating NICE (Narrow Band Imaging International Colorectal Endoscopic classification) Type 1 or Type 2 colorectal polyps. The treatment will typically be carried out under sedation. Small risks for this procedure include complications such as bleeding, intestinal perforation, infection and an adverse reaction to the anaesthetic medication. Patients who have been treated with electroporation have also reported the following symptoms following treatment: pyrexia, obstipation, diarrhea, pyrexia, nausea, headaches, and joint pain. Patients will be required to return for the first follow-up visit, approximately 6 weeks after the initial treatment, at which time they will need to have a colonoscopy. If there is evidence that the initial treatment has not removed 100% of the polyp, an additional treatment will be offered, or the polyp will be removed by Endoscopic Mucosal Resection (EMR) which is the standard treatment for this indication. This decision will be taken by the patient's primary physician. Patients who have an additional treatment will return approximately 12 weeks after the initial treatment for another colonoscopy that falls outside of standard of care protocol. All other visits fall under the standard care timelines. Patients who have successfully been treated with endoscopic ablation will undergo a biopsy at either the first, or second follow up visit to exclude residual disease. This will be performed when the patient is under sedation

Clinical review and colonoscopy will be repeated at 6weeks, 6months and 5years from initial contact to assess the effectiveness on the polyp and the safety of the patient

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age.
* Ability to review the consent form prior to enrolment into the study • Patients must be mentally capable of understanding the information given • Patients must give written informed consent prior to undergoing any study-specific procedures.
* Patients must have at least one polyp (treatment naive, recurrent or residual) measuring >5mm, located distal to the splenic flexure(i.e descending colon, Sigmoid colon, recto sigmoid junction and the rectum above the dentate line)
* Polyp(s) must be classified as Type 1 or Type 2, based on NICE (Narrow Band Imaging International Colorectal Endoscopic) classification; OR Type 1 or Type 2A based on JNET (Japan Narrow Band Imaging Expert Team) classification
* Patients must have a World Health Organization (WHO) performance status ≤ 2 . Patients must have a life expectancy of at least 6 months

Exclusion Criteria:

* < 18 years of age.
* Patients who are incapacitated, unconscious or from a vulnerable population. • Patient who is pregnant or breastfeeding
* Patients unable to provide their own informed consent
* Patients with complex / challenging polyp(s), including but not limited to those that are: o >20mm in size o Flat/bulky in shape o Extending beyond 2 haustra folds or occupying more than 1/3rd of the lumenal circumference o Located on the right colon proximal to the splenic flexure, ileocecal valve, hepatic and splenic flexure or dentate line of the rectum o Fibrosis from large lateral spreading lesions
* Patients with NICE Type 3 category polyps, OR JNET Type 2B or Type 3 polyps
* Patients with British Society of Gastroenterology (BSG) category C (high risk polyps).
* Five or more polyps in a single patient
* Grossly inflamed colonic mucosa with bleeding or ulcers
* Implanted colonic stents
* Polyposis syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consenting adults with endoscopically confirmed colorectal polyps who fit the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Month 6
  Safety evaluation will be performed using reported adverse events (AE) according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
  Treatment emergent AEs include intraprocedural and delayed perforation, bleeding and pain.

SECONDARY OUTCOMES:
Efficacy of pulsed field ablation in the treatment of colorectal polyps | Week 6, Month 6
  Efficacy will be assessed by reviewing the number of polyps that require retreatment following the initial PFA treatment. Images obtained during standard colonoscopies will be used for this assessment.
Efficacy of pulsed field ablation in the treatment of colorectal polyps | Week 6, Month 6
  The amount of polyp(s) removed (in percentage)
Efficacy of pulsed field ablation in the treatment of colorectal polyps | Week 6, Week 12, Month 6, Month12, Month 36, Month 60
  The rate of recurrence of colorectal polyp (in percentage)
Efficacy of pulsed field ablation in the treatment of colorectal polyps | Week 6, Month 6
  The number of polyp(s) treated per session (in numerical value)
Efficacy of pulsed field ablation in the treatment of colorectal polyps | Week 6, Month 6
  The time required for each session of treatment (in seconds)
Efficacy of pulsed field ablation in the treatment of colorectal polyps | Week 6, Month 6
  The 'non-lifting sign' for fibrosis (either present or absent)
Evaluation of Quality of Life following pulsed field ablation treatment of colorectal polyps | Baseline, Week 6, Week 12, Month 6, Month 12, Month 36, Month 60
  Change in Quality of Life Patient Reported Outcomes as measured by Short Form 12 (SF-12) Questionnaire. The scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.